CLINICAL TRIAL: NCT00018512
Title: Biological Specifications for Denture Designs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURG-030-99S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Tooth Loss
Keywords: dental implant
MeSH Terms: conditions — Tooth Loss | interventions — Dental Prosthesis, Implant-Supported

INTERVENTIONS:
Procedure: Implant-supported denture

SUMMARY:
The primary term goal of these research efforts has been to enhance the functional status, comfort and quality of life of edentulous patients by evaluating clinical procedures, denture designs and adjunctive therapies based upon a clear understanding of: (1) oral functional impairments caused by the loss of teeth and subsequent tissue changes; (2) neurophysiological mechanisms associated with oral functions; (3) metabolism of oral tissues; and (4) interactions between biological and psychological processes and denture characteristics. The primary purpose of the proposed clinical outcome study is to compare the relative efficacies of three different combinations of implant-supported maxillary and mandibular prostheses with traditional complete dentures for edentulous patients. Completion of this study will determine the relative cost-effectiveness of the implant-supported denture treatments for use in the general population of edentulous patients.

ELIGIBILITY:
Inclusion criteria:

* Completely edentulous veterans with clinically acceptable conventional dentures.
* Both male and female applicants will be accepted and the prospective participants will be from 35 to 80 years of age.
* Patients who have been completely edentulous for at least two years and have clinically acceptable conventional dentures, which have been worn for at least 6 months.

Exclusion criteria:

* Verified history of medical conditions such as connective tissue disorders, blood dyscrasias, uncontrolled endocrine disorders, active tuberculosis, AIDS, leukemias, Hodgkins, liver disfunction, osteoporosis, chronic nephritis, any chronic condition with life expectancy of less than five years as well as patients on long-term steroids, anticoagulants, and radiation therapy.
* Extremely poor oral hygiene. Oral hygiene condition will be assessed from the amount of food debris, plaque and calculus in their present dentures.
* Insufficient mandibular or maxillary bone height to accommodate 10 mm long implants in potential implant sites.
* Presence of temporomandibular joint dysfunction and evidence of severe bruxism.
* Physician determines a contraindication for oral surgery.
* Candidate expresses reservations about participating for at least three years.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States